CLINICAL TRIAL: NCT06152354
Title: Efficacy of Pediatric Rotary File System Versus Hand Instrumentation for Root Canal Preparation in Primary Teeth: An In Vivo and In Vitro Study
Brief Title: Efficacy of Pediatric Rotary File System Versus Hand Instrumentation for Root Canal Preparation in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 124/2018
Record Dates: First submitted 2023-10-29; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2022-10

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 20 mandibular primary molars in which pulpectomy were performed by hand instrumentation system using K- File from size 15 to size 35.
  Interventions: Device: Manual files
- Experimental group (Experimental): 20 mandibular primary molars in which pulpectomy were performed by rotary system using Kedo-SG rotary file system according to manufacturer's instructions .
  Interventions: Device: rotary system

INTERVENTIONS:
Device: rotary system — crown down technique using Kedo-SG file rotary system using endodontic motor
  Other Names: rotary files
  Arms: Experimental group
Device: Manual files — instrumentation were done by step back technique using K- file (Mani ) from size 15 to size 35 in quarter pull turn motion apically
  Other Names: hand instrumentation
  Arms: Control group

SUMMARY:
The teeth were randomly allocated in two equal groups :

Control group (A):- included 20 mandibular primary molars in which pulpectomy were performed by hand instrumentation system using K- File from size 15 to size 35.

Experimental Group (B):- included 20 mandibular primary molars in which pulpectomy were performed by rotary system using Kedo-SG rotary file system according to manufacturer's instructions

Methods of Evaluation

Stage I :- During and after canal preparation:- The following parameters were evaluated for all cases in both groups:- A- The instrumentation and canal filling time were recorded for both groups using stopwatch. B- Radiographic assessment for filling were done immediately postoperative to record :-

1. Distance between the apex to filling level of the mesial and distal roots .
2. Obturation form

Stage II : Follow up :

The follow up were carried out by clinical and radiographic evaluation for all cases in both groups:-

The clinical evaluation were carried out at (0 base line = after 7 days ) then after 1 , 3 , 6 and 12 months .

Radiographic evaluation were performed immediately postoperative as (0 baseline ) after cementation of stainless steel crowns for assessment of filling quality. Radiographs will be used for comparison for consequent radiographs . Follow ups were performed after 6 and 12 months.

DETAILED DESCRIPTION:
The planned study is a randomized clinical controlled trial including apparently healthy children who were selected from the patients attending the Out- Patient Clinic , Pediatric Dentistry Department, Faculty of Dentistry, Suez Canal University. Informed written consent were obtained from parents or guardians of the children after full explanation of clinical procedures and detailed treatment plan.

The teeth were randomly allocated in two equal groups :

Control group (A):- included 20 mandibular primary molars in which pulpectomy were performed by hand instrumentation system using K- File from size 15 to size 35.

Experimental Group (B):- included 20 mandibular primary molars in which pulpectomy were performed by rotary system using Kedo-SG rotary file system according to manufacturer's instructions

Clinical procedures :

1. Preoperative digital periapical radiograph were taken using standardized paralleling technique using XCP device .
2. Local anesthesia were administered to the patient.
3. The tooth were isolated using rubber dam .
4. Caries were removed by large spoon excavator.
5. The cavities were cleaned by thoroughly rinsing with chlorohexidine 0.2% .
6. Access cavity were done under constant water cooling and suction using high speed round bur No.330 .
7. Pulp chamber were completely deroofed .
8. No .10 size K file were used to determine patency of canals.
9. The working length were determined by apex locator & periapical radiograph.
10. Depending on the group allocation , the canal instrumentation were done by step back technique using K- file (Mani ) from size 15 to size 35 in quarter pull turn motion apically or by crown down technique using Kedo-SG file rotary system using endodontic motor.

11 - After each instrumentation , the canal were irrigated by 1% sodium hypochlorite .

12- The canal were dried with paper points( #30 &#35) 13- Then canal were filled with creamy mix of Zinc oxide & Egenol. 14-Zinc phosphate cement were placed over Zinc oxide & Egenol then finally restored by Stainless steel crown .

15-Postoperative digital periapical radiographs were taken using standardized paralleling technique using XCP device .

Methods of Evaluation

Stage I :- During and after canal preparation:- The following parameters were evaluated for all cases in both groups:- A- The instrumentation and canal filling time were recorded for both groups using stopwatch. B- Radiographic assessment for filling were done immediately postoperative to record :-

1. Distance between the apex to filling level of the mesial and distal roots .
2. Obturation form

Stage II : Follow up :

The follow up were carried out by clinical and radiographic evaluation for all cases in both groups:-

The clinical evaluation were carried out at (0 base line = after 7 days ) then after 1 , 3 , 6 and 12 months .

The following clinical criteria were evaluated: -

* Spontaneous pain as described by Oginin and Undoye ( 29)
* Sensitivity to percussion presence or absence.
* Tooth mobility presence or absence.
* Examination of any changes of the mucobuccal folds (presence or absence of swelling, sinus, draining fistula or abscess).

If the tooth exhibits any of above clinical features, the pulpectomy was considered a failure (F); otherwise, it was regarded as clinical success (S).

Radiographic evaluation were performed immediately postoperative as (0 baseline ) after cementation of stainless steel crowns for assessment of filling quality. Radiographs will be used for comparison for consequent radiographs . Follow ups were performed after 6 and 12 months.

The following radiographic criteria were evaluated :-

* Presence or absence of widening of apical periodontal membrane space .
* Presence or absence of furcation radioluency .
* Presence or absence of internal or external root resorption .

All patients were examined using standardized intra oral paralleling periapical direct digital radiographs using the rinn (XCP) periapical film holder and a long cone. Radiometric and radiodensitometric analysis of the radiographs were carried out using the software of Digora (2.5) system.

Dates of follow up visits were written on the patient 's recall card , parents were asked to call if any symptoms of pain or infection occurred at any time before recall visit .If there is any complications during follow up periods, different techniques of treatment were done according to the case.

ELIGIBILITY:
Inclusion Criteria:

mandibular primary molars with deep caries indicated for pulpectomy

* Restorable lower primary molars.
* History of spontaneous pain or pain that is not relieved by analgesics.
* Pain with percussion
* Excessive bleeding from the root canals

Exclusion Criteria:

* Allergy to any medications used .
* Inability to come in recall visits . mandibular primary molars with exclusion criteria as follows:-
* Acute or chronic abscess & fistula.
* Inter-radicular or periapical bone destruction (radiolucency) as revealed in the preoperative periapical radiograph .
* Mobility grade III.
* Internal root resorption.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Spontaneous Pain | baseline (immediately after procedure), after 7 days, after 1 month, 3 months, 6 months and 12 months from baseline
  A scale from 1 to 10 where 1 is mild pain and 10 Worst pain
Sensitivity to percussion | baseline (immediately after procedure), after 7 days, after 1 month, 3 months, 6 months and 12 months from baseline
  Presence (1) or Absence (0)
Tooth mobility | baseline (immediately after procedure), after 6 months and 12 months from baseline
  Presence (1) or absence (0)
Changes in mucobuccal folds (swelling, abscess or fistula) | baseline (immediately after procedure), after 7 days, after 1 month, 3 months, 6 months and 12 months from baseline
  Presence (1) or Absence (0)
Radiographic examination " internal or external root resorption" | baseline (immediately after procedure), after 6 months and 12 months from baseline
  Presence (1) or absence (0)
Radiographic examination " furcation radiolucency" | baseline (immediately after procedure), after 6 months and 12 months from baseline
  Presence (1) or absence (0)
Radiographic evaluation " widening of apical periodontal membrane space " | baseline (immediately after procedure), after 6 months and 12 months from baseline
  Presence (1) or absence (0)

SECONDARY OUTCOMES:
The instrumentation and canal filling time | immediately postoperative
  recorded for both groups using stopwatch
Radiographic assessment | immediately postoperative
  Distance between the apex to filling level of the mesial and distal roots . Obturation form

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No